CLINICAL TRIAL: NCT04051619
Title: Oxytocin to Reduce Stress-induced Craving in Individuals With Opioid Use Disorder
Brief Title: Oxytocin, Stress, Craving, Opioid Use Disorder
Acronym: OSCO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Carolina L Haass-Koffler, Associate Professor, Brown University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1904002426; P20GM130414 (NIH)
Record Dates: First submitted 2019-08-06; First posted 2019-08-09 (Actual); Results first posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oxytocin first, then placebo (Experimental): Oxytocin was administered as 40 IU/0.12 mL nasal spray in each nostril once in the morning and once in the afternoon for 7 days. After a 2 day washout period, Placebo was administered as nasal spray in each nostril once in the morning and once in the afternoon for 7 days.
  Interventions: Drug: intranasal oxytocin, 40 IU, twice a day for 7 days
- Matching placebo, then oxytocin (Placebo Comparator): Placebo was administered as nasal spray in each nostril once in the morning and once in the afternoon for 7 days. After a 2 day washout period, oxytocin was administered as 40 IU/0.12 mL nasal spray in each nostril once in the morning and once in the afternoon for 7 days.
  Interventions: Drug: intranasal oxytocin, 40 IU, twice a day for 7 days

INTERVENTIONS:
Drug: intranasal oxytocin, 40 IU, twice a day for 7 days — Adjunct therapy
  Other Names: Pitocin

SUMMARY:
Although stress has long been linked to substance use, craving and relapse, there are no available medications that target stress-induced substance use disorder (SUD). In particular, with the rise in opioid use, there is still a crucial need for developing effective pharmacological treatments that target and integrate the complexity of this disease. The long term goal of this project is to identify the key neuroendocrine pathways that are responsible for stress-induced craving in individuals with opioid use disorder (OUD) in order to better understand how they can be effectively treated.

DETAILED DESCRIPTION:
The goal of this research is to evaluate whether oxytocin, a hormone with anti-stress properties, dampens the effects of stress and opioid-associated cues on opioid craving and thus may be an effective adjunctive treatment for OUD.

The central hypothesis of this research is that oxytocin will reduce stress-induced opioid craving in patients with OUD treated with buprenorphine/naloxone as opioid replacement therapy (ORT). This hypothesis is based on the model of addiction (Koob, Neuron 2008) in which chronic substance use and stress lead to neurobehavioral counter-adaptations that dysregulate biobehavioral response.

In this double-blind, cross-over, placebo controlled, randomized trial, individuals with OUD (N=20 who are currently receiving treatment with buprenorphine/naloxone or methadone will be randomized to intranasal oxytocin (40 international units, IU) and oxytocin-matched placebo, administered twice/day for 7 days with a minimum of two days between the opposite condition (oxytocin or placebo). On days 5 and 7, and on days 14 and 16, participants will complete two counter-balanced sessions in which they receive yohimbine (32.4 mg) or yohimbine-matched placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male or female (50%), 18 to 70 (inclusive) years of age;
* Currently meets DSM-5 criteria for OUD;
* Currently on a stable dose of buprenorphine/naloxone or methadone for at least 3 months;
* In good health as confirmed by medical history, physical examination and blood work (Liver function within 5x the Upper normal limits (AST/ALT) and renal function within 2x the Lower Normal Limit (bilirubin, creatine clearance).
* Willing to take medication and adhere to the study procedures;- Understand informed consent and questionnaires in English at an 8th grade level;
* Clinical Opiate Withdrawal Scale (COWS) = 0 at study screening and prior laboratory sessions.

Exclusion Criteria:

* Women who are breastfeeding, test positive for pregnancy or are unwilling to use medically-approved birth control;
* Suicide attempts in the last three months;
* Current substance disorder other than marijuana, nicotine and caffeine as assessed by self-report and urine toxicology screen at baseline;
* Current use of medications that may interact with study medications;
* History of hypersensitivity to study medications;
* Clinically significant electrolyte abnormalities, current rhinitis or use of vasoconstricting medications or prostaglandins.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2023-12-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Brown University, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Gully BJ, Brown ZE, Hornbacher R, Brown JC, Back SE, McCance-Katz EF, Swift RM, Haass-Koffler CL. Oxytocin Reduces Noradrenergic-Induced Opioid-Like Withdrawal Symptoms in Individuals on Opioid Agonist Therapy. Biol Psychiatry Glob Open Sci. 2024 Sep 18;5(1):100395. doi: 10.1016/j.bpsgos.2024.100395. eCollection 2025 Jan. PMID 39534517

RESULTS

PARTICIPANT FLOW:
Groups:
- Oxytocin First, Then Placebo: Oxytocin was administered as 40 IU/0.12 mL nasal spray in each nostril once in the morning and once in the afternoon for 7 days: Adjunct therapy
- Matching Placebo First, Then Oxytocin: Placebo was administered as nasal spray in each nostril once in the morning and once in the afternoon for 7 days: Adjunct therapy
Period: 1st Allocation, 7 Days
Arm/Group | Oxytocin First, Then Placebo | Matching Placebo First, Then Oxytocin
Started (Participants began the first arm of intervention in crossover design, receiving either oxytocin or placebo for 7 days. Between days 5-7 of this arm of the intervention, participants completed 2 laboratory sessions (Visit 3 and 4) under a randomized stress induction procedure (yohimbine) and a matched placebo (yohimbine-placebo). These administrations were counter balanced.) | 10 | 10
Received Yohimbine and Matched Placebo During Lab Sessions 3 and 4. (4 participants were withheld the yohimbine and matched-yohimbine-placebo during lab sessions for safety reasons. These participants completed the sessions under naturalistic conditions with no stress induction.) | 8 | 8
Completed | 10 | 10
Not Completed | 0 | 0
Period: 2nd Allocation (Cross Over)
Arm/Group | Oxytocin First, Then Placebo | Matching Placebo First, Then Oxytocin
Started (Participants began the second arm of intervention in crossover design, receiving the opposite condition to that which they received (oxytocin or matched placebo) for 7 days. Between days 5-7 of this arm of the intervention, participants completed 2 identical laboratory sessions to that of the first arm (Visit 5 and 6) under an identical randomized stress induction procedure (yohimbine and matched placebo).) | 10 (Participants (n=2) enrolled in between-subject design prior COVID-19 did not have the crossover condition. Participant (n=2) was lost at follow up) | 10 (Participants (n=2) enrolled in between-subject design prior COVID-19 did not have the crossover condition. Participant (n=1) was lost at follow up)
Received Yohimbine and Matched Placebo During Lab Sessions 5 and 6. (3 participants were withheld the yohimbine and matched-yohimbine-placebo during lab sessions 5 and 6 for safety reasons. These participants completed the sessions under naturalistic conditions with no stress induction.) | 5 | 5
Completed | 7 | 6
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 1 | 2
Not completed — Completed the study prior to initiation cross-over design | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Outcome measures are grouped into a single arm: all study participants. This is because the crossover design led participants to receive both oxytocin and the matched placebo during the study.
Arm/Group | All Study Participants
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.6 (11.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black or multiracial | 4
  Race: Caucasian | 16
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20
Clinical Opiate Withdrawal Scale (COWS) [Mean (Standard Deviation); unit: score on an 11-item scale] | .9 (1.4)

OUTCOME MEASURES:

1. Primary Outcome: Opioid Craving
Description: The primary outcome will test the effect of oxytocin, compared to placebo, on opioid craving during two laboratory stress induction, paired to a cue reactivity paradigm. The dependent measure for the primary aim is the Desire for Drug Questionnaire (DDQ). The stress induction will be done using yohimbine or matching placebo (counterbalanced) during the two laboratory sessions.
  At each visit the DDQ will be administered 3 times: before starting any procedure, after the yohimbine challenge, and after the cue-reactivity. This outcome will be compared between oxytocin and matching-placebo.
  Minimum score=0 no craving at all, maximum score= 91 severe craving (13 questions on a 7-step Likert-scale)
Time Frame: Before starting any procedure, after the yohimbine challenge, and after the cue-reactivity at each laboratory session, which occurred between days 5-7 and days 14-16.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Oxytocin: Oxytocin was administered as 40 IU/0.12 mL nasal spray in each nostril once in the morning and once in the afternoon for 7 days: Adjunct therapy
- Matching Placebo: Placebo was administered as nasal spray in each nostril once in the morning and once in the afternoon for 7 days.
Arm/Group | Oxytocin | Matching Placebo
Number analyzed (Participants) | 16 | 17
score on a scale
  baseline (yohimbine condition) | 21.6 (7.55) | 22.4 (6.26)
  after stress (yohimbine condition) | 23.3 (7.66) | 23.4 (7.53)
  cue exposure (yohimbine condition) | 22.9 (8.09) | 23.0 (7.92)
  baseline (yohimbine-placebo condition) | 22.7 (7.85) | 19.5 (6.16)
  after stress (yohimbine-placebo condition) | 23.1 (6.95) | 21.7 (7.18)
  cue exposure (yohimbine-placebo condition) | 22.6 (6.74) | 20.9 (7.88)

2. Secondary Outcome: Safety and Tolerability of Oxytocin and Yohimbine in OUD Individuals Receiving Opioid Agonist Therapy: Opiate Withdrawal Syndrome
Description: Participants will complete a laboratory session that includes a battery of medical/physiological/psychological assessments to monitor adverse events. Safety measures include: opiate withdrawal syndrome by Clinical Opiate Withdrawal Scale (COWS) pre and post the laboratory procedures. The COWS is an 11-item scale designed to be administered by a clinician. Minimum=0 (no withdrawal); Maximum=36 (sever withdrawal). The stress induction will be done using yohimbine or matching placebo (counterbalanced) during the two laboratory sessions. High score worse outcome.
  At each visit the COWS will be administered 2 times: before starting any procedure, and after the cue-reactivity. This outcome will be compared between oxytocin and matching-placebo.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxytocin | Matching Placebo
Number analyzed (Participants) | 16 | 17
score on a scale
  Baseline (Yohimbine Condition) | 1.2 (1.17) | 0.8 (.75)
  Post (Yohimbine Condition) | 1.8 (2.23) | 3.0 (3.30)
  Baseline (Yohimbine-placebo Condition) | 1.0 (1.45) | 1.3 (1.38)
  Post (Yohimbine-placebo Condition) | 0.7 (0.84) | 0.6 (1.10)

3. Secondary Outcome: Safety and Tolerability of Oxytocin and Yohimbine in OUD Individuals Receiving Opioid Agonist Therapy: Anxiety
Description: Participants will complete a laboratory session that includes a battery of medical/physiological/psychological assessments to monitor adverse events. Safety measures include: monitor anxiety (HAMA) during lab sessions. Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of Minimum=0 (not present), Maximum=56 (sever), where <17 mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe. The stress induction will be done using yohimbine or matching placebo (counterbalanced) during the two laboratory sessions. High score worse outcome.
  At each visit the HAMA will be administered 3 times: before starting any procedure, after the yohimbine challenge, and after the cue-reactivity. This outcome will be compared between oxytocin and matching-placebo.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Matching Placebo: Placebo was administered as nasal spray in each nostril once in the morning and once in the afternoon for 7 days.: Adjunct therapy
Arm/Group | Oxytocin | Matching Placebo
Number analyzed (Participants) | 16 | 17
score on a scale
  Baseline (Yohimbine condition) | 1.8 (2.10) | 2.5 (2.39)
  after stress (Yohimbine condition) | 2.0 (2.98) | 2.7 (3.65)
  after cue exposure (Yohimbine condition) | 1.9 (1.85) | 2.7 (2.53)
  Baseline (Yohimbine-placebo condition) | 1.3 (1.69) | 2.2 (2.35)
  after stress (Yohimbine-placebo condition) | 0.9 (1.3) | 1.2 (1.50)
  after cue exposure (Yohimbine-placebo condition) | 0.9 (1.7) | 1.0 (2.14)

4. Secondary Outcome: Safety and Tolerability of Oxytocin and Yohimbine in OUD Individuals Receiving Opioid Agonist Therapy: Systolic Blood Pressure (SBP)
Description: Participants will complete a laboratory session that includes a battery of medical/physiological/psychological assessments to monitor adverse events. Safety measures include: monitor systolic blood pressure (SBP) during lab sessions. The stress induction will be done using yohimbine or matching placebo (counterbalanced) during the two laboratory sessions.
  At each visit the SBP will be administered 3 times: before starting any procedure, after the yohimbine challenge, and after the cue-reactivity. This outcome will be compared between oxytocin and matching-placebo.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Oxytocin | Matching Placebo
Number analyzed (Participants) | 16 | 17
mmHg
  baseline (yohimbine condition) | 127.9 (19.97) | 124.2 (19.80)
  after stress (yohimbine condition) | 134.2 (21.90) | 137.2 (18.30)
  after cue exposure (yohimbine condition) | 133.4 (28.80) | 147.2 (25.40)
  baseline (yohimbine-placebo condition) | 129.2 (16.30) | 126.9 (20.50)
  after stress (yohimbine-placebo condition) | 120.8 (10.90) | 121.3 (16.60)
  after cue exposure (yohimbine-placebo condition) | 123.9 (16.50) | 123.0 (13.40)

5. Secondary Outcome: Safety and Tolerability of Oxytocin and Yohimbine in OUD Individuals Receiving Opioid Agonist Therapy: Heart Rate (HR)
Description: Participants will complete a laboratory session that includes a battery of medical/physiological/psychological assessments to monitor adverse events. Safety measures include: monitor Heart rate (HR) during lab sessions. The stress induction will be done using yohimbine or matching placebo (counterbalanced) during the two laboratory sessions.
  At each visit the HR will be administered 3 times: before starting any procedure, after the yohimbine challenge, and after the cue-reactivity. This outcome will be compared between oxytocin and matching-placebo.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: beat/min
Groups:
- Matching Placebo: Placebo was administered as nasal spray in each nostril once in the morning and once in the afternoon for 7 days: Adjunct therapy
Arm/Group | Oxytocin | Matching Placebo
Number analyzed (Participants) | 16 | 17
beat/min
  baseline (yohimbine condition) | 83.0 (16.7) | 80.0 (13.9)
  after stress (yohimbine condition) | 75.5 (14.6) | 83.1 (11.2)
  after cue exposure (yohimbine condition) | 74.6 (18.2) | 77.5 (13.1)
  baseline (yohimbine-placebo condition) | 77.9 (16.1) | 80.0 (13.1)
  after stress (yohimbine-placebo condition) | 69.4 (14.7) | 81.0 (12.9)
  after cue exposure (yohimbine-placebo condition) | 66.3 (12.4) | 82.0 (17.9)

6. Other Pre Specified Outcome: Stress-related Response in OUD Individuals Receiving Opioid Agonist Therapy: Salivary Cortisol
Description: Cortisol (biomarker for stress level) will be measured at the same 3 time points as other measures. The stress induction will be done using yohimbine or matching placebo (counterbalanced) during the two laboratory sessions.
  At each visit the cortisol will be administered 3 times: before starting any procedure, after the yohimbine challenge, and after the cue-reactivity. This outcome will be compared between oxytocin and matching-placebo.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ug/dL
Arm/Group | Oxytocin | Matching Placebo
Number analyzed (Participants) | 16 | 17
ug/dL
  baseline (yohimbine condition) | 0.33 (0.15) | 0.24 (0.14)
  after stress (yohimbine condition) | 0.29 (0.11) | 0.27 (0.16)
  after cue exposure (yohimbine condition) | 0.32 (0.25) | 0.80 (0.70)
  baseline (yohimbine-placebo condition) | 0.28 (0.21) | 0.31 (0.31)
  after stress (yohimbine-placebo condition) | 0.23 (0.13) | 0.24 (0.21)
  after cue exposure (yohimbine-placebo condition) | 0.20 (0.11) | 0.17 (0.13)

ADVERSE EVENTS:
Time Frame: Safety and tolerability were measured retrospectively during the one-week outpatient setting
Description: We did not enroll any participant who was at risk of mortality, suicide or serious adverse event
Arm/Group | Oxytocin | Matching Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17
Other Adverse Events (participants affected / at risk) | 8/16 | 8/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxytocin (N=16) | Matching Placebo (N=17)
Dizziness (Nervous system disorders) | 2 (2) | 3 (4)
Decrease in appetite (Gastrointestinal disorders) | 3 (5) | 3 (3)
Difficulty sleeping (Nervous system disorders) | 5 (6) | 6 (6)
Slowness, sleepiness, or fatigue (Nervous system disorders) | 3 (5) | 4 (6)
Difficulty with concentration or attention (Nervous system disorders) | 6 (7) | 3 (4)
Tingling in fingers or toes (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
Tremor (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 3 (5)
Headache (Nervous system disorders) | 3 (5) | 6 (6)
Nervousness or anxiety (Psychiatric disorders) | 7 (12) | 8 (14)
Irritability (Nervous system disorders) | 4 (4) | 3 (3)
Depression or other mood disturbance (Psychiatric disorders) | 8 (9) | 8 (8)
Muscle aches (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)

LIMITATIONS AND CAVEATS:
Attempting to probe and measure opioid craving in this setting. This study utilized a guided opioid visualization technique, the presence of drug paraphernalia, and an opioid-related video cue. These cues were broad, and different aspects of them may have proved significant to participants at different times. While this is a laboratory procedure limitation, it may also further support the use of OAT for craving management. The study's small sample size and balance between males/females.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-05-05): https://cdn.clinicaltrials.gov/large-docs/19/NCT04051619/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-05): https://cdn.clinicaltrials.gov/large-docs/19/NCT04051619/SAP_001.pdf
  • Informed Consent Form (2022-05-05): https://cdn.clinicaltrials.gov/large-docs/19/NCT04051619/ICF_002.pdf